CLINICAL TRIAL: NCT03011437
Title: Diagnosis Ability of Linked Color Imaging for Helicobacter Pylori Infection Compared With White Light Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kashgar 1st People's Hospital (Other)
Responsible Party: Principal Investigator, Bai Yang, Director, Kashgar 1st People's Hospital
Other Study IDs: 2016A020212007
Record Dates: First submitted 2016-12-28; First posted 2017-01-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Helicobacter Pylori Infection
Keywords: linked color imaging; Helicobacter Pylori
MeSH Terms: interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — gastric mucosa
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- cases: Patients who undergo esophagogastroduodenoscopy during 01/12/2016 and 31/12/2016 in the First People's Hospital of Kashgar Region.
  Interventions: Other: Esophagogastroduodenoscopy

INTERVENTIONS:
Other: Esophagogastroduodenoscopy — Esophagogastroduodenoscopy is an examining method for upper gastrointestinal disease.

SUMMARY:
There are lack of endoscopic criteria for diagnosing Helicobacter pylori (H. pylori) infection by conventional white light imaging (WLI). Linked color imaging (LCI) is a newly developed endoscopy technique, which can diagnose mucosal lesions and H. pylori infection by enhancing color contrast of the mucosa. The aim of the study is to investigate the ability of LCI for diagnosing H. pylori infection compared with WLI.

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) is one of the most common chronic bacterial infections in man. And it is the causative factor for peptic ulcer and regarded as a class I carcinogen for gastric adenocarcinoma. Therefore, accurate detection of infection is crucial for devising proper eradication regimens and preventing the more severe GI complications. Detection of H. pylori in the gastric mucosa can be performed via (1) direct detection of the bacterium; culture, histology and polymerase chain reaction or (2) indirect detection of its enzymatic products particularly urease and serum H. pylori-specific antibody examinations. The direct detection methods are complicated and time-consuming. While the indirect detection methods are less accurate. With the wide use of endoscopy, diagnosis of H. pylori infection by endoscopy should be more accurate and easily available. However, there are still lack of endoscopic criteria for diagnosing H. pylori infection by conventional white light imaging (WLI), which correlates poorly with histopathological findings of H. pylori-induced gastritis . The newly modified LCI system (FUJIFILM Co.) can obtain clear and bright endoscopic images by using short-wavelength narrow-band laser light combined with white laser light. LCI technique can enhance the color of the endoscopic images by digital processing, which makes red regions seem redder and white regions seem whiter. Therefore, LCI may facilitate the detection of certain kinds of gastric lesions. As the common thinking, H. pylori-associated gastritis regions are redder than normal mucosa under WLI because of hyperemia following inflammation. And such redness can be enhanced by LCI. However, there is no criterion for this estimating. Red, green and blue (RGB) color model is a basic component system of the hue, of which each color is a composition of different proportions. Thus, the color obtained by endoscopic images can be quantified by RGB model. The study aimed at comparing the ability of WLI and LCI for diagnosing H. pylori infection by using RGB color model and investigating objective and quantifiable endoscopic criteria for predicting H. pylori infection.

ELIGIBILITY:
Inclusion Criteria:

* People who undergo esophagogastroduodenoscopy for possible upper gastrointestinal disease

Exclusion Criteria:

* Patients who have taken proton pump inhibitor, antibiotics, non-steroidal anti-inflammatory drugs, bismuth agent, H2-receptor inhibitor and medicines that can affect the test of H. pylori infection in a month
* Patients with severe systematic disorders
* Patients with accurate gastrointestinal bleeding in a week
* Patients with histories of gastric surgery
* Pregnant and lactating women
* Patients with poor coagulation function
* Patients diagnosed with gastric cancer

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People who undergo esophagogastroduodenoscopy in the First People's Hospital of Kashgar Region. All patients provided written informed consents to undergo esophagogastroduodenoscopy and participate in this study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy, specificity and sensitivity of LCI for diagnosing Hp infection compared with the pathology | one month

SECONDARY OUTCOMES:
Hp infection rate | one month

CONTACTS AND LOCATIONS:
Overall Officials: Zou X Guang, Study Chair — First People's Hospital of Kashgar Region
Locations (1):
- First People's Hospital of Kashgar Region, Kashgar, Xinjiang, China

IPD SHARING:
Plan to Share IPD: No